CLINICAL TRIAL: NCT02827318
Title: Eating Disinhibition and Vagal Tone Moderate the Postprandial Response to Glycaemic Load: A Randomised Controlled Trial
Brief Title: Eating Disinhibition and Vagal Tone and the Postprandial Response to Glycaemic Load
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Principal Investigator, Dr Hayley Young, Dr, Swansea University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DisGL
Record Dates: First submitted 2016-06-29; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Hunger
Keywords: Blood glucose
MeSH Terms: interventions — isomaltulose; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 75g glucose (Active Comparator): 75g of glucose dissolved in 500ml provided in a clear plastic tumbler.
  Interventions: Dietary Supplement: Glucose
- 75g isomaltulose (Experimental): 75g of isomaltulose dissolved in 500ml provided in a clear plastic tumbler.
  Interventions: Dietary Supplement: Isomaltulose
- Sweetened water (Placebo Comparator): 500ml water sweetened with sucralose provided in a clear plastic tumbler.
  Interventions: Dietary Supplement: Sweetened water

INTERVENTIONS:
Dietary Supplement: Isomaltulose — 75g Isomaltulose (low glycaemic load intervention)
  Arms: 75g isomaltulose
Dietary Supplement: Glucose — 75g Glucose (high glycaemic load intervention)
  Arms: 75g glucose
Dietary Supplement: Sweetened water — Sweetened water will be used as a control
  Arms: Sweetened water

SUMMARY:
Reducing the glycaemic load (GL) of the diet may benefit appetite control but its utility is complicated by psychological influences on eating. Disinhibited behaviour, a risk factor for overconsumption, is characterized by reduced prefrontal cortex activity, which in turn directly modulates vagal tone; a phenomenon inversely associated with blood glucose (BG) and insulin levels. This double blind randomised controlled trial explores the influence of disinhibited eating and vagal tone (heart rate variability) on the postprandial response to GL and hunger.

DETAILED DESCRIPTION:
There is growing recognition that lowering the glycaemic load of the diet might reduce a range of cardiovascular risk factors such as raised plasma triglycerides, HbA1c and C reactive protein and aid in body weight regulation. A proposed mechanism includes higher satiety and prolonged satiation by virtue of improved postprandial metabolic control, although, whether lower GL meals result in greater weight loss or increased satiety is still a matter of debate. One matter complicating the issue is that the desire to consume food may be driven by psychological factors; food reward centres in the brain may override hormonal regulation of food intake. Amongst psychological factors disinhibition has the largest and most consistent body of empirical data that associates it with weight gain although the mechanisms involved are unknown. This study will investigate whether, irrespective of BMI or habitual diet, disinhibited eaters have greater glycaemic excursions following a high glycaemic load drink and whether this predicts subsequent satiation.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy adults who scored either high or low on the Three factor eating questionnaire disinhibition subscale

Exclusion Criteria:

Participants were excluded if they

* had a cardiovascular or metabolic disorder
* gastrointestinal problems
* were pregnant
* had a current diagnosis of a mood or eating disorder
* and/or were taking medications or herbal supplements to manage body weight or control appetite

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose | From baseline to 30 minutes
  Blood glucose was monitored from finger pricks using an ExacTech sensor (Medisense Britain Limited) that using an enzymic method, coupled with microelectronic measurement. Change in blood glucose from baseline to after 30 minutes will assess the speed of incline.
Change in blood glucose | from 30 to 150minutes
  As above to assess the speed of decline.

SECONDARY OUTCOMES:
Hunger | 30, 150 minutes
  Participants were asked to respond to the question "how hungry are you feeling right now" on a single 100mm visual analogue scale anchored by "Not at all" and "Extremely".

CONTACTS AND LOCATIONS:
Locations (1):
- Swansea University, Swansea, West Glamorgan, United Kingdom

REFERENCES:
- [Derived] Young HA, Watkins H. Eating disinhibition and vagal tone moderate the postprandial response to glycemic load: a randomised controlled trial. Sci Rep. 2016 Oct 20;6:35740. doi: 10.1038/srep35740. PMID 27761024